CLINICAL TRIAL: NCT05671107
Title: Development and Validation of an Online Neurobehavioral Evaluation Tool for PTEN Hamartoma Tumor Syndrome (PHTS)
Brief Title: Development and Validation of an Online Neurobehavioral Evaluation Tool for PTEN Patients
Status: Completed | Type: Observational
Sponsor: John Carroll University (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-013; JCU-20-001 (Other Grant/Funding Number: PTEN Research Foundation)
Record Dates: First submitted 2022-12-16; First posted 2023-01-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: PTEN Hamartoma Tumor Syndrome
Keywords: Neurodevelopmental disorders; PTEN; PHTS; Autism; Online Assessment; Neurobehavioral
MeSH Terms: conditions — Hamartoma Syndrome, Multiple; Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PTEN - with NDD: Patients diagnosed with PTEN Hamartoma Tumor Syndrome and a neurodevelopmental disorder including but not limited to autism spectrum disorder, attention-deficit disorder / attention-deficit hyperactivity disorder, speech language disorder(s), intellectual disability, global developmental delay, oppositional defiant disorder, and / or motor or developmental disorders.
  Interventions: Diagnostic Test: NET
- PTEN - without NDD: Patients diagnosed with PTEN Hamartoma Tumor Syndrome
  Interventions: Diagnostic Test: NET
- Sibling Controls: Siblings related to patients with diagnosis of PTEN Hamartoma Tumor Syndrome
  Interventions: Diagnostic Test: NET
- Unrelated Controls: Unrelated participants with no known genetic or neurodevelopmental disorder
  Interventions: Diagnostic Test: NET

INTERVENTIONS:
Diagnostic Test: NET — Online survey measuring a variety of developmental domains including anxiety, motor, daily living skills, challenging behaviors, social communication, restrictive and repetitive behaviors, ADHD, executive functioning, mood, quality of life, and sleep

SUMMARY:
The purpose of this study is to develop a survey completed by parents, caregivers, or other informants that evaluates several important domains of functioning relevant to individuals with neurodevelopmental disorders, including autism spectrum disorder and people with genetic syndromes. Participation in this research will include assisting the research team in the development of the survey measures.

DETAILED DESCRIPTION:
With greater understanding of the biology of PTEN Hamartoma Tumor Syndrome (PHTS), including patients with and without neurodevelopmental disorder (NDD) phenotypes, there is potential to develop novel personalized therapeutics. Given the recent observation that many PHTS patients with and without NDD have significant neurobehavioral manifestations, it will be crucial to broadly track a range of neurobehavioral domains as part of future trials. Unfortunately, there are few well-validated measures that would be appropriate for the full range of presentations in the PHTS population. Further, as a rare genetic syndrome, PHTS patients are geographically distributed making frequent data collection during research very difficult. Thus, the overarching aim of this proposal is to develop and validate an online neurobehavioral evaluation tool (NET) with caregiver-report survey scales and patient-completed webcam-collected performance measures that captures key neurobehavioral information. In partnership with patients, caregivers, and scientist-clinician experts, the study will develop, pilot test, and validate NET survey and performance measures. Specifically, at least 240 caregiver-patient pairs will be recruited (patient ages 4-24) from PHTS without NDD, PHTS with NDD, and controls (sibling and unrelated healthy controls). NET data will be collected at baseline, 1-month, and 4-month follow-up. Aim 1 will focus on the development and validation of brief, psychometrically-sound NET survey scales. Aim 2 will conduct group comparisons on NET measures. Aim 3 will use longitudinal data to evaluate short-term stability of NET survey scales and describe neurobehavioral change within and across study groups. The project will also explore the feasibility of performance measure collection, provide initial psychometric evaluation, and conduct a group comparison of performance measures. If the project aims are achieved, and future validation supports research and clinical use, the NET will be an efficient, reliable, valid, co-normed, multi-modal instrument, that, by virtue of online (at-home) administration, will decrease patient and family burden and increase the temporal resolution and power of future longitudinal studies and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Has a PTEN Hamartoma Tumor Syndrome diagnosis with or without a neurodevelopment disorder
* Access to a tablet (10+ inch screen), laptop, or desktop computer
* Access to reliable internet
* Able to attend to short videos (30 plus seconds)
* Able to hear audio from a computer device
* Able to see without corrective lenses

Ages: 3 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Social Communication Interaction | Baseline
  Develop survey questions and scales related content areas for Social Communication Interactions. Social communication refers to the emergence of verbal and nonverbal skills, social interaction, and social cognition
Social Communication Interaction | One month follow up
  Develop survey questions and scales related content areas for Social Communication Interactions. Social communication refers to the emergence of verbal and nonverbal skills, social interaction, and social cognition
Social Communication Interaction | Four month follow up
  Develop survey questions and scales related content areas for Social Communication Interactions. Social communication refers to the emergence of verbal and nonverbal skills, social interaction, and social cognition
Daily Living Skills | Baseline
  Develop questions and survey scales related to content areas of activities of daily living. Activities of daily living are activities related to personal care. They include bathing or showering, dressing, getting in and out of bed or a chair, walking, using the toilet, and eating.
Daily Living Skills | One month follow up
  Develop questions and survey scales related to content areas of activities of daily living. Activities of daily living are activities related to personal care. They include bathing or showering, dressing, getting in and out of bed or a chair, walking, using the toilet, and eating.
Daily Living Skills | Four months later
  Develop questions and survey scales related to content areas of activities of daily living. Activities of daily living are activities related to personal care. They include bathing or showering, dressing, getting in and out of bed or a chair, walking, using the toilet, and eating.

SECONDARY OUTCOMES:
Restrictive and Repetitive Behaviors | Baseline
  Develop survey and rating scales related to content areas for restrictive and repetitive behaviors. Restricted and repetitive behaviors and interests are among the three core symptoms of autism. They include repetitive movements with objects, repeated body movements such as rocking and hand-flapping, ritualistic behavior, sensory sensitivities and circumscribed interests
Restrictive and Repetitive Behaviors | One month follow up
  Develop survey and rating scales related to content areas for restrictive and repetitive behaviors. Restricted and repetitive behaviors and interests are among the three core symptoms of autism. They include repetitive movements with objects, repeated body movements such as rocking and hand-flapping, ritualistic behavior, sensory sensitivities and circumscribed interests
Restrictive and Repetitive Behaviors | Four month follow up
  Develop survey and rating scales related to content areas for restrictive and repetitive behaviors. Restricted and repetitive behaviors and interests are among the three core symptoms of autism. They include repetitive movements with objects, repeated body movements such as rocking and hand-flapping, ritualistic behavior, sensory sensitivities and circumscribed interests
Anxiety | Baseline
  Develop survey questions and scales related to content areas for anxiety. Anxiety is what we feel when we are worried, tense or afraid - particularly about things that are about to happen, or which we think could happen in the future
Anxiety | One month follow up
  Develop survey questions and scales related to content areas for anxiety. Anxiety is what we feel when we are worried, tense or afraid - particularly about things that are about to happen, or which we think could happen in the future
Anxiety | Four month follow up
  Develop survey questions and scales related to content areas for anxiety. Anxiety is what we feel when we are worried, tense or afraid - particularly about things that are about to happen, or which we think could happen in the future
Motor Skills | Baseline
  Develop survey questions and scales related to content areas for motor skills.A motor skill is a function that involves specific movements of the body's muscles to perform a certain task. These tasks could include walking, running, or riding a bike. In order to perform this skill, the body's nervous system, muscles, and brain have
Motor Skills | One month follow up
  Develop survey questions and scales related to content areas for motor skills.A motor skill is a function that involves specific movements of the body's muscles to perform a certain task. These tasks could include walking, running, or riding a bike. In order to perform this skill, the body's nervous system, muscles, and brain have
Motor Skills | Four month follow up
  Develop survey questions and scales related to content areas for motor skills.A motor skill is a function that involves specific movements of the body's muscles to perform a certain task. These tasks could include walking, running, or riding a bike. In order to perform this skill, the body's nervous system, muscles, and brain have
Challenging Behaviors | Baseline
  Develop survey questions and rating scales related to content areas for challenging behaviors.A person's behaviour can be defined as "challenging" if it puts them or those around them (such as their carer) at risk, or leads to a poorer quality of life. It can also impact their ability to join in everyday activities. Challenging behaviour can include: aggression. self-harm.
Challenging Behaviors | One month follow up
  Develop survey questions and rating scales related to content areas for challenging behaviors.A person's behaviour can be defined as "challenging" if it puts them or those around them (such as their carer) at risk, or leads to a poorer quality of life. It can also impact their ability to join in everyday activities. Challenging behaviour can include: aggression. self-harm.
Challenging Behaviors | Four month follow up
  Develop survey questions and rating scales related to content areas for challenging behaviors.A person's behaviour can be defined as "challenging" if it puts them or those around them (such as their carer) at risk, or leads to a poorer quality of life. It can also impact their ability to join in everyday activities. Challenging behaviour can include: aggression. self-harm.
ADHD | Baseline
  Develop survey questions and rating scales related to content areas for ADHD. Refers to the ongoing pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or development.
ADHD | One month follow up
  Develop survey questions and rating scales related to content areas for ADHD. Refers to the ongoing pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or development.
ADHD | Four month follow up
  Develop survey questions and rating scales related to content areas for ADHD. Refers to the ongoing pattern of inattention and/or hyperactivity-impulsivity that interferes with functioning or development.
Executive Functioning | Baseline
  Develop survey questions and rating scales related to content areas for executive functioning. Executive functioning and self-regulation skills are the mental processes that enable us to plan, focus attention, remember instructions, and juggle multiple tasks successfully.
Executive Functioning | One month follow up
  Develop survey questions and rating scales related to content areas for executive functioning. Executive functioning and self-regulation skills are the mental processes that enable us to plan, focus attention, remember instructions, and juggle multiple tasks successfully.
Executive Functioning | Four month follow up
  Develop survey questions and rating scales related to content areas for executive functioning. Executive functioning and self-regulation skills are the mental processes that enable us to plan, focus attention, remember instructions, and juggle multiple tasks successfully.
Mood | Baseline
  Develop survey questions and rating scales related to content areas for mood. Focusing on particular feelings or a state of mind.
Mood | One month follow up
  Develop survey questions and rating scales related to content areas for mood. Focusing on particular feelings or a state of mind.
Mood | Four month follow up
  Develop survey questions and rating scales related to content areas for mood. Focusing on particular feelings or a state of mind.
Quality of Life | Baseline
  Develop survey questions and rating scales related to content areas for quality of life including family, financial, etc.
Quality of Life | One month follow up
  Develop survey questions and rating scales related to content areas for quality of life including family, financial, etc.
Quality of Life | Four month follow up
  Develop survey questions and rating scales related to content areas for quality of life including family, financial, etc.
Sleep | Baseline
  Develop survey questions and rating scales related to content areas for sleep patterns and behaviors.
Sleep | One month follow up
  Develop survey questions and rating scales related to content areas for sleep patterns and behaviors.
Sleep | Four month follow up
  Develop survey questions and rating scales related to content areas for sleep patterns and behaviors.

CONTACTS AND LOCATIONS:
Locations (2):
- John Carroll Univeristy, University Heights, Ohio, United States
- University Hospital South Hampton, Hampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan to upload deidentified data to Open Science Framework
Supporting Information: CSR
Time Frame: Within one year of study completion
URL: https://osf.io/cguzs/